CLINICAL TRIAL: NCT06628804
Title: Effects of Artemisia and Green Tea Extracts on Promoting Gastric Mucosal Health in Adults With Functional Dyspepsia: A Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Artemisia and Green Tea Extracts for Gastric Mucosal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 12-2024-006
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Functional Dysphonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artemisia and green tea extracts group (Experimental): This group takes Artemisia and green tea extracts for 8 weeks.
  Interventions: Dietary Supplement: Artemisia and green tea extracts
- Placebo group (Placebo Comparator): This group takes a placebo for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Artemisia and green tea extracts — Artemisia and green tea extracts 700 mg/day for 8 weeks
  Arms: Artemisia and green tea extracts group
Dietary Supplement: Placebo — Placebo 700 mg/day for 8 weeks
  Arms: Placebo group

SUMMARY:
This clinical trial aims to determine whether Artemisia and green tea extracts promote gastric mucosal health in adults with functional dyspepsia and to assess its safety.

The main questions are:

* Does Artemisia and green tea extracts promote gastric mucosal health in participants?
* What side effects occur when participants take Artemisia and green tea extracts?

DETAILED DESCRIPTION:
Researchers will compare Artemisia and green tea extracts to placebo to evaluate their effectiveness in promoting gastric mucosal health.

Participants will:

* Take Artemisia and green tea extracts or a placebo daily for 8 weeks.
* Visit the clinic every 4 weeks for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* Rome IV-based functional dyspepsia-

Exclusion Criteria:

* Patients with gastrointestinal symptoms requiring immediate drug treatment.
* Individuals with a history of hypersecretory gastric disorders like Zollinger-Ellison syndrome.
* Individuals who received Helicobacter pylori eradication therapy within 4 weeks prior to the trial.
* Individuals who have taken nonsteroidal anti-inflammatory drugs, steroids, antibiotics, aspirin, antithrombotic agents, or acid suppressants within the last month.
* Individuals with a history of upper gastrointestinal surgery, stricture, bleeding, or procedures like esophageal dilation or mucosal resection within the last year.
* Individuals with gastric ulcers (active or healing), duodenal ulcers (active or healing), reflux esophagitis (LA grade A or higher), or malignant tumors identified within the last 6 months through endoscopy.
* Patients with uncontrolled hypertension (resting BP ≥160/100 mmHg).
* Patients with uncontrolled diabetes (fasting glucose ≥160 mg/dL).
* Individuals with creatinine levels ≥ 2 times the upper limit of normal at the research institution.
* Individuals with aspartate aminotransferase or alanine aminotransferase levels ≥ 2 times the upper limit of normal at the research institution.
* Alcohol abusers.
* Individuals taking medications for psychiatric disorders (except those taking intermittent medication for sleep disorders).
* Pregnant or breastfeeding women or those planning to become pregnant during the clinical trial period.
* Individuals with allergies to any components of the study foods.
* Individuals who participated in or plan to participate in another drug clinical trial within the last month.
* Individuals deemed unsuitable for the study by the investigator for other reasons.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
The Korean version of the Gastrointestinal Symptom Rating Scale: Total score | From enrollment to the end of treatment at 8 weeks
  Measured at baseline and 8 weeks. This is a 4-point Likert scale for each of the 15 items, with scores ranging from 0 to 3. A score of 0 indicates no symptoms, and 3 represents very severe symptoms. The higher the overall score, the more severe the gastrointestinal symptoms. The minimum value was 0, and the maximum value was 45, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The Korean version of the Gastrointestinal Symptom Rating Scale: Subtotal scores of upper abdomen | From enrollment to the end of treatment at 8 weeks
  Measured at baseline and 8 weeks. This is a 4-point Likert scale for each of the 8 items, with scores ranging from 0 to 3. A score of 0 indicates no symptoms, and 3 represents very severe symptoms. The higher the overall score, the more severe the gastrointestinal symptoms. The minimum value was 0, and the maximum value was 21, and higher scores mean a worse outcome.
Visual Analogue Scale for evaluating gastric mucosal improvement | From enrollment to the end of treatment at 8 weeks
  Measured at baseline and 8 weeks. The minimum value was 0 and the maximum value was 100, and higher scores mean a worse outcome.
Gastrointestinal symptom score | From enrollment to the end of treatment at 8 weeks
  Measured at baseline and 8 weeks. The minimum value was 0 and the maximum value was 40, and higher scores mean a worse outcome. For each gastrointestinal symptom, the minimum value was 0, and the maximum value was 4, and higher scores mean a worse outcome.
Patient's global assessment score | From enrollment to the end of treatment at 8 weeks
  Measured at baseline and 8 weeks. The 5-point Likert scale for the Patient's Global Assessment Score is a self-reported tool where patients rate their disease activity. It uses an order scale, with 5 indicating "Very Good" and 1 indicating "Poor." The patient evaluates their condition based on this scale: Very Good-Good-Fair-Unchanged-Poor.
Pepsinogen I level (ng/mL) | From enrollment to the end of treatment at 8 weeks
  Measured at baseline and 8 weeks
Pepsinogen II level (ng/mL) | From enrollment to the end of treatment at 8 weeks
  Measured at baseline and 8 weeks
Pepsinogen I/Pepsinogen II ratio | From enrollment to the end of treatment at 8 weeks
  Measured at baseline and 8 weeks
Gastrin-17 level (ng/L) | From enrollment to the end of treatment at 8 weeks
  Measured at baseline and 8 weeks
Helicobacter pylori IgG titer (units) | From enrollment to the end of treatment at 8 weeks
  Measured at baseline and 8 weeks
High-sensitive C-reactive protein (mg/dL) | From enrollment to the end of treatment at 8 weeks
  Measured at baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD,PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea